CLINICAL TRIAL: NCT05438225
Title: Automated Text Message Reminders to Promote Hearing Healthcare Access - Pilot Study
Brief Title: Text Message Reminders for Hearing Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Uchechukwu Megwalu, Associate Professor of Otolaryngology - Head & Neck Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-66347
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Hearing Loss
Keywords: hearing loss; elderly; primary care; text message
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated Text Message Reminder (Experimental): Participants will receive automated reminder text instructing them to discuss hearing issues with their PCPs, and to request a referral to audiology or otolaryngology if they have hearing loss.
  Interventions: Behavioral: Automated text message reminder
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Automated text message reminder — Participants in the intervention group will receive monthly automated reminder text instructing them to discuss hearing issues with their PCPs, and to request a referral to audiology or otolaryngology if they have hearing loss.
  Arms: Automated Text Message Reminder

SUMMARY:
Many individuals with hearing loss do not receive adequate hearing healthcare. Given their close and long-term relationships with patients, primary care providers (PCPs) could play a vital role in improving access to hearing healthcare. Unfortunately, hearing loss is often underdiagnosed in primary care settings, because hearing screening is not a routine part of primary care visits, and the responsibility often falls on the patient or family to recognize and address the issue. The investigators propose to pilot test the use of text message reminders to encourage elderly patients to discuss hearing assessment with there PCPs. The study objectives are to: 1) design an automated text-messaging reminder system; 2) assess the feasibility of deploying the intervention in a clinical trial setting; and 3) evaluate whether the intervention increases willingness to seek hearing healthcare.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult patients aged 65 and older
* Have not audiometric testing within the past 5 years
* Has had at least one prior visit encounter with a Stanford primary care provider the past 1 year
* Has a cell phone with a valid phone number

Exclusion Criteria:

* History of childhood hearing loss
* Hearing aid users
* Limited English proficiency

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Likelihood of patient-physician discussion of hearing loss or hearing assessment | 3 months after enrollment
  Participant-reported rating of the likelihood of discussing hearing assessment with their PCP in the next 6 months. Likelihood will be assessed on an 11-point visual analogue scale (VAS). Score range: 0 to 10 (0 = not likely, 10 = very likely). Participants who have already discussed hearing assessment with their PCP will be assigned a score of 10.

SECONDARY OUTCOMES:
Likelihood of obtaining audiogram | 3 months after enrollment
  Participant-reported rating of the likelihood of obtaining an audiogram in the next 6 months. Likelihood will be assessed on an 11-point visual analogue scale (VAS). Score range: 0 to 10 (0 = not likely, 10 = very likely). Participants who have already undergone audiometric testing will be assigned a score of 10.
Likelihood of obtaining hearing aids | 3 months after enrollment
  Participant-reported rating of the likelihood of obtaining hearing aids if an audiogram showed significant hearing loss. Likelihood will be assessed on an 11-point visual analogue scale (VAS). Score range: 0 to 10 (0 = not likely, 10 = very likely). Participants who have already obtained hearing aids will be assigned a score of 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No